CLINICAL TRIAL: NCT07025239
Title: A Randomized, Double-blind, Multicenter Phase 3 Study of QL1706 Injection in Combination With Bevacizumab and XELOX Versus Placebo in Combination With Bevacizumab and XELOX as First-line Therapy for the Treatment of Patients With Unresectable Metastatic Colorectal Cancer (mCRC)
Brief Title: QL1706 Injection Plus Bevacizumab and XELOX vs Placebo Plus Bevacizumab and XELOX as First-Line Treatment of Unresectable Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL1706-309
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 + bevacizumab + XELOX (Experimental)
  Interventions: Drug: QL1706; Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine
- Placebo+ bevacizumab + XELOX (Placebo Comparator)
  Interventions: Drug: Bevacizumab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Placebo

INTERVENTIONS:
Drug: QL1706 — QL1706 will be administered by IV infusion at 5mg/kg on Day 1 of each 21-day cycle until disease progression (PD), intolerable toxicity, initiation of a new anti-tumor therapy, death, withdrawal of informed consent, loss to follow-up or other conditions requiring termination of the treatment (whichever occurs first). The administration of QL1706 lasts for up to 2 years.
  Arms: QL1706 + bevacizumab + XELOX
Drug: Bevacizumab — Bevacizumab will be administered by IV infusion at 7.5mg/kg on Day 1 of each 21-day cycle until disease progression (PD), intolerable toxicity, initiation of a new anti-tumor therapy, death, withdrawal of informed consent, loss to follow-up or other conditions requiring termination of the treatment (whichever occurs first). The administration of Bevacizumab lasts for up to 2 years.
Drug: Oxaliplatin — Oxaliplatin will be administered by IV infusion at 130 mg/m2 on Day 1 of each 21-day cycle up to 8 treatment cycles.
Drug: Capecitabine — Capecitabine will be administered orally at 1000 mg/m2 twice daily for 2 consecutive weeks, followed by one-week rest in each 21-day cycle until disease progression (PD), intolerable toxicity, initiation of a new anti-tumor therapy, death, withdrawal of informed consent, loss to follow-up or other conditions requiring termination of the treatment (whichever occurs first). The administration of Capecitabine lasts for up to 2 years.
Drug: Placebo — Placebo will be administered by IV infusion at 5mg/kg on Day 1 of each 21-day cycle until disease progression (PD), intolerable toxicity, initiation of a new anti-tumor therapy, death, withdrawal of informed consent, loss to follow-up or other conditions requiring termination of the treatment (whichever occurs first). The administration of Placebo lasts for up to 2 years.
  Arms: Placebo+ bevacizumab + XELOX

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of QL1706 Injection in combination with bevacizumab and XELOX compared with placebo in combination with bevacizumab and XELOX for first-line treatment in patients with unresectable mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily sign the informed consent form (ICF) and can understand and comply with the study requirements;
* Males and females aged 18 to 75 years old (including boundary value) on the date of signing ICF;
* Unresectable metastatic colorectal adenocarcinoma confirmed by histopathology examination;
* No previous systemic anti-tumor drug therapy for metastatic colorectal adenocarcinoma;
* At least one target lesion as judged by the investigator per RECIST v1.1 (lesions previously treated with topical treatment such as radiotherapy should not be considered as target lesions, unless it is confirmed that there has been definite progression of lesions located in the previous radiotherapy region);
* Be able to provide sufficient previously archived tumor tissue samples or agree to collect tumor tissue samples (≥ 5 unstained pathological tissue sections) by biopsy for biomarker testing. If sufficient tissue samples cannot be provided, it should be determined with the sponsor;
* ECOG PS score of 0 or 1 within 7 days before the first dose;
* Adequate liver, bone marrow, and renal organ function.

Exclusion Criteria:

* Patients had other active malignant tumors within 5 years prior to the first dose. Patients with localized tumors that have been cured, such as basal cell carcinoma of the skin, squamous cell carcinoma of skin, superficial bladder carcinoma, carcinoma in situ of prostate, cervical carcinoma in situ, and breast carcinoma in situ, can be enrolled.
* Previous treatment with radiotherapy at any site within 4 weeks prior to the first dose.
* Previous treatment with postoperative adjuvant therapy with targeted drugs targeting epidermal growth factor receptor (EGFR), vascular endothelial growth factor (VEGF) or its receptor (VEGFR), including but not limited to Bevacizumab, Cetuximab, Panitumumab, Aflibercept, Regorafenib or Anlotinib;
* Previous treatment with any T cell costimulation or immune checkpoint inhibitors, including but not limited to anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4, anti-OX-40 or anti-CD137 monoclonal antibodies;
* Participation in a clinical study and treatment with study drug or device within 4 weeks prior to the first dose, or traditional Chinese medicine treatment < 2 weeks from the first dose;
* Patients who have a history of severe (≥ Grade 3) gastrointestinal ulcers, gastrointestinal perforation, fistula formation, intra-abdominal inflammation/abscess, intra-abdominal pneumatosis not due to puncture or surgery, macroscopic digestive tract hemorrhage/melena (excluding hemorrhoidal hemorrhage), and hemoptysis (about 3 mL or more) within 6 months prior to the first dose;
* Uncontrollable pleural effusion, pericardial effusion or ascites requiring drainage;
* Presence of dysphagia and unable to swallow the investigational product;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) Assessed by the Independent Radiology Review Committee (IRRC) | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented progressive disease or deaths (whichever comes first), assessed per RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 66 months
  OS is defined as the time from the randomization to deaths, regardless of the cause of deaths
Progression Free Survival (PFS) Assessed by Investigator | Up to approximately 2 years
  OS is defined as the time from the randomization to deaths, regardless of the cause of deaths
Objective Response Rate (ORR) | Approximately 36 months
  ORR is defined as the proportion of subjects who achieve a best response of complete response (CR) or partial response (PR) per RECIST v1.1 criteria
Duration Of Response (DOR) | Approximately 36 months
  ORR is defined as the proportion of subjects who achieve a best response of complete response (CR) or partial response (PR) per RECIST v1.1 criteria
Incidence of AEs, SAEs and treatment-emergent adverse events (TEAEs). | From the subject signs the ICF to 30 days after the last dose of study drug is administered
  Adverse events (AEs), serious adverse events (SAEs), treatment-emergent adverse events are included. The investigator should carry out judgment for investigational drug correlation